CLINICAL TRIAL: NCT00097071
Title: Safety and Efficacy of Insulin Aspart Versus Insulin Lispro in Insulin Pumps in Children and Adolescents With Type 1 Diabetes
Brief Title: Safety and Efficacy of NovoLog vs. Humalog in Insulin Pumps in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-2181
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Diabetes, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin lispro
Drug: insulin aspart

SUMMARY:
This trial is conducted in the United States of America (USA). It is demonstrated that intensive insulin therapy resulting in good glycaemic control can reduce or delay the incidence of complications secondary to Type 1 Diabetes. Insulin Aspart (NovoLog®) is an ideal insulin to use in an intensive insulin regimen using continuous subcutaneous insulin injection (CSII) therapy in the pediatric and adolescent age population. This trial compares the safety and efficacy of Insulin Aspart (NovoLog®) and Insulin Lispro (Humalog®) delivered by CSII in children and adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 299 (Actual)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 16 weeks treatment

SECONDARY OUTCOMES:
Measurements of glycaemic control, safety parameters including frequency of hypoglycaemia, laboratory tests, clinical evaluations and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (47):
- United States (47):
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Loma Linda, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Englewood, Colorado
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Hackensack, New Jersey
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Manhasset, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Charleston, West Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Weinzimer SA, Ternand C, Howard C, Chang CT, Becker DJ, Laffel LM; Insulin Aspart Pediatric Pump Study Group. A randomized trial comparing continuous subcutaneous insulin infusion of insulin aspart versus insulin lispro in children and adolescents with type 1 diabetes. Diabetes Care. 2008 Feb;31(2):210-5. doi: 10.2337/dc07-1378. Epub 2007 Nov 5. PMID 17989308
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com